CLINICAL TRIAL: NCT04038034
Title: Clinical Evaluation of the Antioxidant and Neuroprotective Effects of CoQ10-MINIACTIVES® (COQUN® OS) 100 mg BID Oral Administration in Patients Affected by Primary Open Angle Glaucoma (POAG): a Randomized, Double Blind Study
Brief Title: Valuation of the Antioxidant and Neuroprotective Effects of CoQ10-MINIACTIVES® (COQUN® OS) in Patients Affected by Primary Open Angle Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VISUfarma SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VF-GLAU-CoQ10/2019
Record Dates: First submitted 2019-05-09; First posted 2019-07-30 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Placebo Comparator): 35 patients treated with pressure lowering drugs and placebo
  Interventions: Dietary Supplement: Placebo
- group B (Experimental): 35 patients with pressure lowering drugs and COQUN oral formulation 100 mg BID.
  Interventions: Dietary Supplement: CoQ10- MINIACTIVES

INTERVENTIONS:
Dietary Supplement: CoQ10- MINIACTIVES — COQUN oral formulation 100 mg BID
  Arms: group B
Dietary Supplement: Placebo — Placebo
  Arms: group A

SUMMARY:
This is a randomized, double blind study with competitive enrolment, aimed to enroll a total of 70 patients with a diagnosis of primary open angle glaucoma (POAG).

Patients, after signing the Informed Consent, will enter into a 1- week screening phase during which the baseline tests will be conducted.

Subjects will be randomized in a 1:1 ratio to the following groups:

* group A of 35 patients treated with pressure lowering drugs and placebo;
* group B of 35 patients with pressure lowering drugs and COQUN oral formulation 100 mg BID.

ELIGIBILITY:
Inclusion criteria:

* Patient Informed consent form (ICF) signed
* M & F Aged ≥ 40 and ≤ 80 years at the time of the signature of ICF
* Patients with Primary Open Angle Glaucoma (POAG) stage early-moderate according to Hodapp-Parrish-Anderson criteria (MD less than -12 dB)
* Patients must be diagnosed with POAG at least 1 year before the screening visit in this study.
* Anamnesis with at least 1 value of Intraocular pressure (IOP) >21mmHg documented any time prior the initiation of the stable treatment with anti-hypertensive topical drugs.
* Patients affected by POAG and under stable treatment with anti-hypertensive topical drugs in the previous 6 months prior to enrolment to maintain IOP ≤18 mmHg.
* Corrected visual acuity (using ETDRS tables) ≥ 8/10
* Transparent dioptric means to allow the examination of the OCT >25 μm.
* Pachymetry values between 500 and 600 μm.
* Patients have to show a stable visual field in the previous 6 months prior to enrolment (where by stable visual field it is intended that the patient must remain within the same stage of POAG severity (i.e. early or moderate) during the previous 6 months before the enrolment).
* Willing to follow all study procedures, including attending all site visits, tests and examinations.
* Women must agree to be using two forms of effective contraception, be post-menopausal from at least 12 months prior to trial entry, or surgically sterile.

Exclusion criteria:

* Patients with a severe defect of POAG according to Hodapp-Parrish-Anderson criteria.
* Previously diagnosed optic neuropathies.
* Diabetic retinopathy or Hypertensive retinopathy.
* Decompensated diabetes.
* Not stabilized hypertension (SAP and/or DAP) despite under adequate pharmacological treatment.
* Retinal pathologies including hereditary forms.
* Neurological, neurodegenerative or cerebrovascular conditions.
* No previous history or presence of any disease involving cornea or retina.
* Patients with a significantly progressive opacity of lens in the previous 3 months prior to enrolment (where by significant progressive opacity of lens it is intended patients who have been diagnosed with cataracts of any aetiology and for whom surgery is being considered).
* No surgical intervention for cataract in the previous 3 months prior to enrolment.
* Eye inflammatory conditions (uveitis) diagnosed any time in the patient's history.
* Treatment with topical or systemic neuroprotective agents different from CoQ10. These patients can be admitted in the study after at least a 1 month of wash-out period.
* Treatment with warfarin.
* Treatment with miotic drugs able to influence the visual field.
* Treatment with systemic or topical steroids.
* Refractive defects beyond the 5 spherical diopters, both positive and negative and over 3 cylindrical.
* Any clinically significant history of serious digestive tract, liver, kidney, cardiovascular, cancer or hematological disease.
* Known drug and/or alcohol abuse.
* Mental incapacity that precludes adequate understanding or cooperation.
* Participation in another investigational study or blood donation within 3 months prior to ICF signature.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Pattern Electroretinogram Amplitude (PERG P50-N95 A) | between the baseline visit (V0) and the last study visit after 12 months of treatment (V3)
  To evaluate the difference of mean changes of Pattern Electroretinogram Amplitude (PERG P50-N95 A) (μV) observed between the two study groups.

SECONDARY OUTCOMES:
Pattern Electroretinogram Amplitude (PERG P50-N95 A) | between the baseline visit (V0) and Month 4 and Month 8 and the last study visit after 12 months of treatment (V3)
  To evaluate the difference of mean changes of Pattern Electroretinogram Amplitude (PERG P50-N95 A) (μV) observed between the two study groups.
Pattern Electroretinogram Amplitude Implicit Times (PERG P50 IT) | between the baseline visit (V0) and Month 4 and Month 8 and the last study visit after 12 months of treatment (V3)
  To evaluate the changes from baseline to each study visit between the two study groups in Pattern Electroretinogram Amplitude Implicit Times (PERG P50 IT) in milliseconds (ms)
Visual Evoked Potentials Implicit Times (VEP P100 IT) | between the baseline visit (V0) and Month 4 and Month 8 and the last study visit after 12 months of treatment (V3)
  To evaluate the changes from baseline to each study visit between the two study groups in Visual Evoked Potentials Implicit Times (VEP P100 IT) in milliseconds (ms)
Visual Evoked Potentials Amplitude (VEP N75-P100 A) | between the baseline visit (V0) and Month 4 and Month 8 and the last study visit after 12 months of treatment (V3)
  To evaluate the changes from baseline to each study visit between the two study groups in Visual Evoked Potentials Amplitude (VEP N75-P100 A) in microvolt (μV)
Visual field | from baseline to each study visit (V1, V2, V3)
  To evaluate the changes from baseline to each study visit between the two study groups in Visual field (separately MD and PSD) evaluated by Humphrey field analyzer (HFA) Sita Standard 30-2
Contrast sensitivity | between the baseline visit (V0) and Month 4 and Month 8 and the last study visit after 12 months of treatment (V3)
  To evaluate the changes from baseline to each study visit between the two study groups in Contrast sensitivity measured with Vistech tables (Vision Chart from CSO)
Optical Coherence Tomography | between the baseline visit (V0) and Month 4 and Month 8 and the last study visit after 12 months of treatment (V3)
  To evaluate the changes from baseline to each study visit between the two study groups in Peripapillary retinal nerve fiber layer (RNFL) thickness, macular RNFL, macular ganglion cell layer (GCL), macular inner plexiform layer (IPL) assessed with natural pupils by the means of spectral domain Optical Coherence Tomography (OCT, Heidelberg Spectralis)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - UO Oculistica - PO Cisanello, Pisa, PI
  - U.O. di Oculistica, Fondazione Policlinico Agostino A. Gemelli,, Rome

IPD SHARING:
Plan to Share IPD: Undecided